CLINICAL TRIAL: NCT01447004
Title: a Case-control Study of the Association Between Heavy Mental and Children With Attention Deficit Hyperactivity Disorder in Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: hushhirb
Record Dates: First submitted 2011-10-04; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Heavy metal has been reported that it can cause attention deficit and behavioral disturbance. The investigators hypothesis is that heavy metal is associated with children with attention deficit/hyperactivity disorder(ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet DSM-IV criteria for ADHD based-on the K-Schedule for affective disorder and schizophrenia(K-SADS-PL-K) interview

  * Subjects signed a written consent form voluntarily.
  * Patient 's assent to participate in the study and written informed consent form signed by one of the parents, parent surrogates, or legal guardian.
  * Subjects/parents, parent surrogates or legal guardian who can understand the participation of the study and voluntarily withdraw from the study at any time

Exclusion Criteria:

* Subjects who have any history of bipolar disorder, psychotic disorder, and substance use disorder, have been diagnosed with a pervasive developmental disorder, organic brain disease and seizure disorder.
* Subjects who have significant suicidal ideation or homicidal ideation
* Subjects with mental retardation
* Subjects with Tourette's syndrome requiring drug therapy.
* Subjects who currently have a significant medical conditions (e.g. diseases of cardiovascular, hepatic, renal, respiratory, glaucoma).
* Subjects who have abnormalities in the ECG or show clinically significant abnormalities of laboratory results, including serum chemistries and hematology.
* Subjects who have been administrated alpha-2 adrenergic receptor agonist,antidepressant, antipsychotic, benzodiazepines, modafinil, anticonvulsant within recent 2 months.
* Subjects who dyed their hair within 8 weeks

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects must meet DSM-IV criteria for ADHD based-on the K-Schedule for affective disorder and schizophrenia(K-SADS-PL-K) interview
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-03

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym university sacred heart hospital, Anyang, Gyeonggi-do, South Korea